CLINICAL TRIAL: NCT03583580
Title: A Multicenter Phase Ⅱ Prospective Clinical Trial of Accelerated Partial Breast Irradiation With IMRT After Breast-conserving Surgery in Early Breast Cancer
Brief Title: Accelerated Partial Breast Irradiation With IMRT in Early Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shulian Wang, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC201804006
Record Dates: First submitted 2018-06-19; First posted 2018-07-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms; Neoplasm Recurrence, Local
Keywords: Breast conserving surgery; Accelerate partial breast irradiation; intensity-modulated radiation therapy; phase II
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Recurrence, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerated Partial Breast Irradiation (Experimental): Accelerated partial breast irradiation (APBI) to the region of tumour bed
  Interventions: Radiation: Accelerated Partial Breast Irradiation

INTERVENTIONS:
Radiation: Accelerated Partial Breast Irradiation — Patients are irradiated to the region of tumour bed using intensity modulated radiation therapy (IMRT)

SUMMARY:
This study is to evaluate the efficacy and toxicity of accelerated partial breast irradiation (ABPI) with intensity modulated radiation therapy (IMRT) in low-risk breast cancer treat with breast-conserving surgery.

DETAILED DESCRIPTION:
This study is a national multicenter phase II prospective clinical trial to enroll low-risk breast cancer treat with breast-conserving surgery. All eligible patients will receive ABPI to a total dose of 40Gy, in 10 fractions, 4Gy/fx/day, within 2 weeks. Intensity modulated radiation therapy (IMRT) technique is used. During Follow up, the locoregional recurrence,survival,acute and late adverse events,and quality of life will be prospectively evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Life Expectation: > 5 years
* Enrollment date no more than 12 weeks after breast-conserving surgery or no more than 8 weeks after adjuvant chemotherapy
* Histologically confirmed diagnosis of invasive ductal carcinoma (grade 1-2), or mucinous carcinoma, or papillary carcinoma, or tubular carcinoma, or medullary carcinoma: primary tumor ≤ 3.0cm in maximum diameter and pN0; or histologically confirmed DCIS: primary tumor ≤ 2.5cm in maximum diameter, low-medium grade
* Unifocal tumour (confirmed by diagnostic MRI)
* No lymphovascular invasion
* ER positive (defined as medium-strongly nuclear staining in >1% of the cancer cells)
* Negative radial resection margins of >= 2 mm
* Surgical clips placed in the tumor bed
* Written informed consent.

Exclusion Criteria:

* Stage Ⅱ-Ⅲ
* Multifocal tumors
* Histologically confirmed diagnosis of invasive ductal carcinoma (grade 3), invasive micropapillary carcinoma, carcinoma of lobular in situ, invasive lobular carcinoma
* Paget's disease of the nipple
* Underwent oncoplastic surgery of ipsilateral breast
* Underwent neoadjuvant chemotherapy or hormonal therapy
* Previous or simultaneous contralateral breast cancer
* Undergone ipsilateral chest wall radiotherapy
* Active collagen vascular disease.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female only
Enrollment: 537 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
locoregional control rate | 5 years
  ipsilateral breast and axilla nodal relapse rate

SECONDARY OUTCOMES:
overall survival | 5 years
  any death
disease-free survival | 5 years
  any recurrence or death
distant-metastasis survival | 5 years
  distant metastasis

OTHER OUTCOMES:
acute and late adverse events assessed by CTCAE v4.0 | 5 years
  acute skin toxicity,breast swelling, breast pain,radiation pneumonitis, cardiac toxicity, pulmonary fibrosis, cosmetic result
quality of life measured with BR-23 questionnaire | 2 years
  BR-23 questionnaire
the incidence of second malignancy | 5 year
  pathologically diagnosis of contralateral breast cancer and other malignant tumors after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Shulian Wang, M.D., Principal Investigator — National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No